CLINICAL TRIAL: NCT03029975
Title: The Influence of Regular Beef Consumption and Protein Density of the Diet on Training-induced Gains in Muscle Strength and Performance in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16997
Record Dates: First submitted 2017-01-19; First posted 2017-01-24 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-08

CONDITIONS: Aging
Keywords: beef; protein; resistance training; strength; performance
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: This study will consist of two groups: one group will be asked to consume 2x the RDA of protein during the 10 week intervention, while the other group will be asked to consume the RDA for protein. Both groups will receive 10 weeks of the same resistance training intervention.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RDA (Active Comparator): Participants will be asked to consume the RDA for protein for a 10 week period while also undergoing progressive resistance training exercise three times a week. Beef protein consumption will be emphasized and participants will consume a beef meal after each training session.
  Interventions: Behavioral: Resistance Training Exercise; Behavioral: Beef Protein Consumption
- 2x RDA (Experimental): Participants will be asked to consume the twice the RDA for protein for a 10 week period while also undergoing progressive resistance training exercise three times a week. Beef protein will be emphasized and participants will consume a beef meal after each training session.
  Interventions: Behavioral: Resistance Training Exercise; Behavioral: Beef Protein Consumption

INTERVENTIONS:
Behavioral: Resistance Training Exercise — Participants will undergo 10 weeks of progressive resistance exercise training while following their randomly assigned nutritional intervention.
Behavioral: Beef Protein Consumption — Following each resistance training sessions, participants will consume either a 3oz or 6oz beef patty (corresponding to the randomly assigned nutritional intervention group). Participants will also be provided with beef protein powder and beef snack bars to help them achieve their assigned protein goals during the intervention period.

SUMMARY:
Humans lose muscle and strength as they get older. Further, ageing is accompanied by loss in cognitive function. It is not quite clear why this happens; however, it is known that the loss of muscle and strength can increase risk for physical and mental health risks and impair the ability of older people to remain physically independent. Weight lifting and proper nutrition, particularly eating high quality protein at the proper time and quantity, may help prevent these losses when a person gets older. To determine if regular beef consumption as part of a higher protein diet aids the muscle adaptive response to resistance training and improvements in cognition, seventy healthy individuals will be recruited to lift weights 3 times a week for 10 weeks. One group (n=36) will consume the Recommended Dietary Allowance (RDA) for protein (0.8g/kg/day), while the other group (n=36) will consume an amount twice the RDA (1.6g/kg/day), which is in agreement with recommendations from the American College of Sports Medicine. Participants will have their muscle strength tested and samples of blood and muscles will be collected before and after training to determine how the muscle adaptive response to resistance exercise is affected by higher protein intake. In addition, participants will undergo cognitive assessments at baseline and follow-up to determine the influence of improving muscle strength on attention and memory. Overall, the investigators proposed study will use sensitive methodology to determine if providing protein above the RDA and at optimal times during the day in combination with a weight lifting program can help make someone stronger and build larger muscles than someone consuming the RDA, as well as what processes may be responsible for helping the muscles to get bigger and stronger.

ELIGIBILITY:
Inclusion Criteria:

* Non-obese adults: BMI <30 kg/m2
* Aged between 40-64 years
* Sedentary
* Weight-stable for 6 months prior

Exclusion Criteria:

* Allergies to beef consumption
* Phenylketonuria (PKU)
* BMI >30 kg/m2
* history of active cardiovascular disease, diabetes mellitus, GI disorders, musculoskeletal/orthopedic disorders (e.g. osteoarthritis, rheumatoid arthritis, tendinitis, gout, fibromyalgia, patellar tendinopathy, or chronic low back pain)
* hypersensitivity or allergy to antibiotics
* Kidney, urinary, or liver conditions
* Epilepsy
* Diagnosed mental illness
* have bleeding or clotting disorders (or take related medications e.g.. Coumadin/ low dose Aspirin)
* High alcohol consumption
* use tobacco
* uncontrolled hypertension
* vegan/vegetarian diets
* on medications known to affect protein metabolism (i.e. corticosteroids, androgen/estrogen containing compounds, non-steroidal anti-inflammatories)
* habitual consumption of high (>1.8 g protein/kg/d) or low (<0.66 g protein/kg/day)
* pregnancy
* supplements that influence protein metabolism (e.g. omega 3 fish oils)

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Maximal strength of leg muscles | Change from baseline to the end of the 10 week diet and resistance training intervention
  Assess maximum strength of legs using an isokinetic dynamometer in combination with 1 repetition maximum testing on leg extension, leg press, and leg curl machines.

SECONDARY OUTCOMES:
Muscle cross-sectional area | Change from baseline to the end of the 10 week diet and resistance training intervention
  Using muscle biopsies, the investigators will assess the muscle cross sectional area of the vastus lateralis pre and post intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Freer Hall, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McKenna CF, Salvador AF, Hughes RL, Scaroni SE, Alamilla RA, Askow AT, Paluska SA, Dilger AC, Holscher HD, De Lisio M, Khan NA, Burd NA. Higher protein intake during resistance training does not potentiate strength, but modulates gut microbiota, in middle-aged adults: a randomized control trial. Am J Physiol Endocrinol Metab. 2021 May 1;320(5):E900-E913. doi: 10.1152/ajpendo.00574.2020. Epub 2021 Mar 8. PMID 33682457